CLINICAL TRIAL: NCT04911478
Title: Long-term Follow-up Protocol for Subjects Treated With Adicet Allogeneic Gamma Delta (γδ) CAR T Cell Investigational Products
Brief Title: Long-term Follow-up Study of Allogeneic Gamma Delta (γδ) CAR T Cells
Status: Enrolling by invitation | Type: Observational
Sponsor: Adicet Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ADI-20200102
Record Dates: First submitted 2021-05-23; First posted 2021-06-03 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Lymphoma, Follicular; Lymphoma, Mantle-Cell; Marginal Zone Lymphoma; Primary Mediastinal B-cell Lymphoma; Diffuse Large B Cell Lymphoma; Lymphoma, Non-Hodgkin
Keywords: B-Cell lymphoma; CAR-T; Cell Therapy; Allogeneic Cell Therapy; T cells gamma delta; Immunotherapy, Adoptive; Antigens, CD20
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Test for RCR following treatment with Adicet Bio allogeneic CAR T cell products. Also will continue to follow immunogenicity assessments of Adicet Bio allogeneic CAR T cell products by using patients blood specimens to assess humoral as well as cellular responses to CAR T cell products. Persistence of ADI-001 will be measured in blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects from Adicet Bio allogeneic γδ CAR T cell interventional studies.: This is a rollover protocol designed to provide long-term follow-up to all subjects previously enrolled in Adicet Bio allogeneic γδ CAR T cell study.
  Patients will be followed for up to 15 years post treatment of Adicet Bio allogeneic γδ CAR T cell investigational products.
  Interventions: Genetic: ADI-001

INTERVENTIONS:
Genetic: ADI-001 — No study drug is administered in this study. Patients who have received Adicet allogeneic γδ CAR T cell therapy will be evaluated in this trial for long-term safety and efficacy

SUMMARY:
The purpose of this study is to assess long-term side effects from subjects who receive an Adicet Bio γδ CAR T cell product. Subjects will join this study once they complete the parent interventional study. No additional study drug will be given, but subjects can receive other therapies for their cancer while they are being followed for long term safety in this study. For a period of 15 years from the first administration of Adicet Bio allogeneic γδ CAR T cell product, subjects will be assessed for long-term safety and survival through collection of data that include safety, efficacy, pharmacokinetics and immunogenicity.

DETAILED DESCRIPTION:
This is a non-therapeutic, multi-center, long-term follow-up (LTFU) study of subjects who received an Adicet Bio allogeneic γδ CAR T cell product that has been genetically engineered to express the anti-CD20 CAR by transduction with a self-inactivating, replication incompetent gamma retroviral vector. The period of follow-up is 15 years after the administration of the γδ CAR T cell product.

The study involves up to 15 years post-infusion monitoring of subjects who have been exposed to a genetically engineered CAR in Adicet Bio clinical studies. Upon early termination/discontinuation or completion of the parent interventional study, subjects will enroll into this study. Collection of these data will further define the risk-benefit and efficacy profile Adicet allogeneic γδ CAR T cell investigational products.

This is an observational study, and the elements of the study design are per published guidelines for gene therapy medicinal products that utilize integrating viral vectors such as gamma retrovirus and it is important to evaluate any delayed adverse events after infusion with such products.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received any Adicet allogeneic CAR T investigational product and have either completed the core treatment protocol or have discontinued early
* All patients who are willing and able to adhere to the study visit schedule and other protocol requirements.
* Capable of giving signed informed consent which includes compliance with requirements and restrictions listed in the informed consent form (ICF) and protocol

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or Female
Study Population: Patients will be enrolled following either the completion or early termination/discontinuation from Study NCT04735471 or any protocol in which patients were administered Adicet allogeneic γδ CAR T cell. Patients will begin the long-term follow-up period regardless of whether they responded to treatment or progressed on treatment. Patients will be followed for up to 15 years post infusion and will continue to be monitored for safety, immunogenicity and efficacy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2038-08 (Estimated); Study Completion 2039-08 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of Adicet Bio allogeneic γδ CAR T cell products | 15 years
  Occurrence of new Adverse Events of Special interests, Serious AEs and malignancies

SECONDARY OUTCOMES:
Measure quantitative immunoglobulin and peripheral blood immunophenotyping | 15 years post last treatment
Monitor for the presence of replication competent retrovirus (RCR) | 15 years post last treatment
  Test for RCR following treatment with Adicet Bio allogeneic γδ CAR T cell products by QCR analysis
Duration of ADI-001 persistence | 15 years post last treatment
  Defined as duration from dosing to undetectable levels of Adicet allogeneic γδ CAR T cell per microliter blood
Overall Response Rate by Lugano Criteria | 15 years post last treatment
  Overall Response Rate by Lugano Criteria
Duration of Response by Lugano Criteria | 15 years post last treatment
  Duration of Response by Lugano Criteria
Progression Free Survival by Lugano Criteria | 15 years post last treatment
  Progression Free Survival by Lugano Criteria
Time To Progression by Lugano Criteria | 15 years post last treatment
  Time To Progression by Lugano Criteria
Overall Survival | 15 years post last treatment
  Overall Survival from date of first treatment until date of death

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Baylor Scott & White Research Institute, Dallas, Texas
  - MD Anderson Caner Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No